CLINICAL TRIAL: NCT03890900
Title: Developing and Evaluating the T2DXcel Mobile Application for Adult Patients With Type 2 Diabetes
Brief Title: T2DXcel Mobile Application
Acronym: T2DXcel
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Sunit P. Jariwala, Associate Professor (Medicine), Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-9590
Record Dates: First submitted 2019-03-23; First posted 2019-03-26 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This proposal will develop, evaluate, and refine a patient-centered mobile application (DiabetesXcel), which will deliver tailored and algorithm-based diabetes education to improve the process and diabetes-related outcomes. We also test the reliability of eHEALS and NVS questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T2DXcel mobile application (Other): T2DXcel is a mobile application (patient-facing) that delivers guideline-based diabetes education.
  Interventions: Other: T2DXcel mobile application

INTERVENTIONS:
Other: T2DXcel mobile application — T2DXcel is a mobile application (patient-facing) that delivers guideline-based diabetes education.

SUMMARY:
Given the need for personalizable and adaptive mobile applications for patients with type 2 diabetes, this proposal will develop, evaluate, and refine a patient-centered mobile application (T2DXcel), which will deliver tailored and algorithm-based diabetes education to improve process and diabetes-related outcomes.

DETAILED DESCRIPTION:
The Bronx has the heaviest burden of diabetes within New York City (NYC) and statewide. The highest diabetes hospitalization and death rates in NYC occur in the Bronx, which has hospitalization rates approximately 25 percent above the statewide average. The Bronx is one of the poorest urban counties in the nation, and diabetes disproportionately impacts high-poverty communities. The borough has an ethnically and racially diverse population (53.5% of residents are Hispanic and 36.5% are black), and diabetes is highly prevalent among blacks and Hispanics. Obesity, a major risk factor for diabetes, is also prevalent with nearly 33% (much higher than the 24% prevalence of obesity in NYC) of Bronx adults being obese. Among the many social determinants of health, medical provider practice behaviors, suboptimal access to health care, lack of patient knowledge regarding proper medication administration and potential side effects, and difficulty adhering to medical regimens by patients and families all contribute to poor diabetes outcomes.

With appropriate medical care including education (especially regarding potentially modifiable lifestyle factors that contribute to diabetes), well-informed patients can achieve diabetes control. However, there are significant challenges in providing effective patient education in the ambulatory setting, such as time constraints and prioritizing other issues (e.g. comorbid conditions) above comprehensive diabetes education. While patient education and teaching self-management skills are critical to improve diabetes outcomes, such strategies will succeed only as part of more comprehensive interventions. Diabetes self-management education (DSME) has been linked to decreases in hemoglobin A1c, reductions in the onset and/or progression of diabetes complications, reductions in diabetes-related hospitalizations and readmissions, and improvements in quality of life, lifestyle behaviors (e.g. physical activity, healthier eating), self-efficacy, and coping skills. The American Association of Diabetes Educators (AADE) has described the AADE7 Self-Care Behaviors (healthy eating, being active, monitoring, taking medications, problem solving, healthy coping, reducing risks) as a framework to organize and structure patient-centered education. Despite the proven benefits of DSME, less than 10% of type 2 diabetes (T2D) patients receive structured education for a variety of reasons: providers' misunderstanding of DSME effectiveness and confusion about how to make referrals; many clinic sites' lack of access to DSME services; and some payers' lack of coverage for DSME services. With the increasing use of smartphones and the internet, health information technology (IT)-based approaches (e.g. mobile applications, text messaging platforms, internet-based educational modules, and telemedicine/telehealth interventions) - through standalone interventions or by supplementing education (i.e. by reinforcing content delivered in-person) - can increase patients' access to DSME, and have been linked to improvements in hemoglobin A1c and other outcomes. Mobile applications ('apps') can provide day-to-day support for patients with diabetes, but commonly lack evidence-based content and/or comprehensiveness. A recent study reported that only a small percentage of the diabetes apps available on the iOS and Android stores supported the AADE7 behaviors regarding problem solving, healthy coping, and reducing risks. Another recent article suggested that few apps provided personalized education or tailored therapeutic support. As with other chronic conditions, diabetes mobile applications are often characterized by low retention rates and decreased user engagement with the app following the initial download.

Given the need for personalizable and adaptive mobile applications for patients with type 2 diabetes, this proposal will develop, evaluate, and refine a patient-centered mobile application (T2DXcel), which will deliver tailored and algorithm-based diabetes education to improve process and diabetes-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

English-speaking individuals >18 years with:

1. T2D (diagnosis made by a healthcare provider) on an anti-diabetic medication with hemoglobin A1c > 6.5% at the time of recruitment and enrollment
2. Diabetes care at Montefiore
3. Able to give informed consent; and d) smartphone (iOS or Android) access

Exclusion Criteria:

1. Pregnancy
2. Chronic illness with organ failure (heart failure, severe liver disease, chronic kidney disease stage 3-4 or dialysis) or requiring chemotherapy or steroid use
3. Severe psychiatric or cognitive problems that would prohibit an individual from completing the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline hemoglobin A1c to 3 and 6 months | Baseline, 3 months, 6 months
  Patients' glycemic control measured by hemoglobin A1c

SECONDARY OUTCOMES:
Patient satisfaction measured by the Client Satisfaction Questionnaire-8 | Baseline, 3 months, 6 months
  Patient satisfaction measured by the Client Satisfaction Questionnaire-8
Change from baseline diabetes knowledge to 3 months and 6 months | Baseline, 3 months, 6 months
  Diabetes knowledge as measured by the validated Diabetes Knowledge Questionnaire-24
Change from baseline diabetes self-management capabilities to 3 months and 6 months | Baseline, 3 months, 6 months
  Diabetes self-management capabilities as measured by the Diabetes Self-Management Questionnaire
Change from baseline diabetes self-efficacy to 3 months and 6 months | Baseline, 3 months, 6 months
  Diabetes self-efficacy as measured by the Diabetes Empowerment Scale-Short Form
Change from baseline diabetes quality of life to 3 months and 6 months | Baseline, 3 months, 6 months
  Patients' diabetes quality of life measured by the Diabetes Quality of Life questionnaire
Change from baseline LDL cholesterol to 3 months and 6 months | Baseline, 3 months, 6 months
  LDL cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Sunit Jariwala, MD, Principal Investigator — Albert Einstein College of Medicine and Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregated and de-identified datasets will be shared with other researchers.